CLINICAL TRIAL: NCT05613751
Title: Enhancing Protection Against Influenza and COVID-19 for Pregnant Women and Medically at Risk Children (EPIC Study)
Brief Title: Enhancing Protection Against Influenza and COVID-19 for Pregnant Women and Medically at Risk Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Helen Marshall, Clinical Research Director, Women's and Children's Health Network Consultant in Vaccinology and Medical Director, Vaccinology and Immunology Research Trials Unit, Women's and Children's Health Network, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: WCHN HREC/2022/HREC00082
Record Dates: First submitted 2022-11-10; First posted 2022-11-14 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Influenza; COVID-19
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Intervention Model Description: Four multi-centre, parallel group, superiority, randomized control trials (with 1:1 allocation) of nudge interventions to improve influenza and COVID-19 vaccine uptake among pregnant women and medically at risk children. Each RCT will enroll 1038 participants (n = 519 each in intervention and control groups), with a total of 4154 participants in the four RCTs:
  * pregnant women's RCTs
    * COVID-19 vaccine (n= 1038): Arm #1 (Standard care, n=519); Arm #2 (Nudge intervention, n=519)
    * Influenza vaccine (n= 1038): Arm #1 (Standard care, n=519); Arm #2 (Nudge intervention, n=519)
  * medically at-risk children's RCTs
    * COVID-19 vaccine (n= 1038): Arm #1 (Standard care, n=519); Arm #2 (Nudge intervention, n=519)
    * Influenza vaccine (n= 1038): Arm #1 (Standard care, n=519); Arm #2 (Nudge intervention, n=519)
  There are eight arms in total for four RCTs.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding is considered desirable; however, it will depend on the type of nudge and will be determined after the nudge is developed. Endpoint measurements will involve low level contact of study staff, however when contact is required (such as AIR/ confirmation of influenza/COVID-19 vaccine receipt etc), this will be carried out by trial staff shielded from information that might reveal trial group assignment. The study statistician undertaking the analysis and study investigators will remain blinded to trial intervention assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Pregnant women-COVID-19 vaccine RCT - intervention group (Experimental): Women randomized to the intervention group will receive the nudge (three text messages four weeks apart) to remind them to get the COVID-19 booster vaccine
  Interventions: Behavioral: Nudge
- Pregnant women-COVID-19 vaccine RCT - standard care group (No Intervention): Women randomized to the standard care group will not receive the nudge (three text messages four weeks apart) to remind them to get the COVID-19 booster vaccine. They will receive normal care at the hospital.
- Pregnant women-influenza vaccine RCT - intervention group (Experimental): Women randomized to the intervention group will receive the nudge (three text messages four weeks apart) to remind them to get the annual influenza vaccine
  Interventions: Behavioral: Nudge
- Pregnant women-influenza vaccine RCT - standard care group (No Intervention): Women randomized to the standard care group will not receive the nudge (three text messages four weeks apart) to remind them to get the annual influenza vaccine. They will receive normal care at the hospital.
- Medically at risk children-COVID-19 vaccine RCT - intervention group (Experimental): Parents of medically at risk children randomized to the intervention group will receive the nudge (three text messages four weeks apart) to remind them to get their child the COVID-19 vaccine
  Interventions: Behavioral: Nudge
- Medically at risk children-COVID-19 vaccine RCT - standard care group (No Intervention): Parents of medically at risk children randomized to the standard care group will not receive the nudge (three text messages four weeks apart) to remind them to get their child the COVID-19 vaccine. They will receive normal care at the hospital.
- Medically at risk children-influenza vaccine RCT - intervention group (Experimental): Parents of medically at risk children randomized to the intervention group will receive the nudge (three text messages four weeks apart) to remind them to get their child the annual influenza vaccine
  Interventions: Behavioral: Nudge
- Medically at risk children-influenza vaccine RCT - standard care group (No Intervention): Parents of medically at risk children randomized to the standard care group will not receive the nudge (three text messages four weeks apart) to remind them to get their child the annual influenza vaccine. They will receive normal care at the hospital.

INTERVENTIONS:
Behavioral: Nudge — Three text messages that are sent four weeks apart reminding to obtain the vaccines
  Arms: Medically at risk children-COVID-19 vaccine RCT - intervention group; Medically at risk children-influenza vaccine RCT - intervention group; Pregnant women-COVID-19 vaccine RCT - intervention group; Pregnant women-influenza vaccine RCT - intervention group

SUMMARY:
Pregnant women and children with chronic medical conditions are at increased risk of hospitalisation, intensive care admission and death from influenza and COVID-19 infections. However, there appears to be a high level of vaccine hesitancy among women of reproductive age. We will develop "nudge" interventions to improve influenza and COVID vaccine uptake and test the effectiveness of the interventions using randomised controlled trials in

* pregnant women
* medically at risk children.

DETAILED DESCRIPTION:
Pregnant women and children with chronic medical conditions are at an unacceptable risk of hospitalisation and death from influenza and COVID-19 infections. Pregnant women are 3 times more likely to die from COVID-19 and over 7 times more likely to be admitted to an intensive care unit (ICU) with influenza compared to non-pregnant women. Children with chronic disease are already compromised with a higher risk of hospitalisation from influenza and requirement for ICU management and long term disability following COVID-19. Uptake of the recommended influenza vaccine among pregnant women and medically at risk children in Australia is only ~50%. Based on recent surveys, the predicted uptake of COVID-19 vaccine among both groups is also likely to be ~50%. These two groups preferentially receive care from medical specialists (obstetricians and paediatricians) and specialist nursing staff in hospitals, and are less likely to engage with primary care, the usual providers of immunisation.

The aim of this project is to develop a nudge (i.e. small changes in the environment that alter people's behaviour) and evaluate the effectiveness of the nudge intervention in improving the uptake of COVID and influenza vaccine by conducting four randomised control trials in

* pregnant women
* medically at risk children.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 pregnant women RCT: Pregnant women have received 2 or less doses of a recommended COVID-19 vaccine
* Influenza pregnant women RCT: Pregnant women have not received the influenza vaccine during pregnancy
* COVID-19 medically at risk children RCT: Medically at risk children aged 5 years to 18 years with a cardiac, endocrine, respiratory, gastrointestinal, haematological, musculoskeletal, neurological condition
* Influenza medically at risk children RCT: Children aged ≥6 months and < 18 years with medical conditions specified in this list: immunocompromising conditions including malignancy, chronic steroid use, haematopoietic stem cell transplant; functional or anatomical asplenia including sickle cell disease or other haemoglobinopathies, congenital or acquired asplenia (for example, splenectomy) or hyposplenia; cardiac disease including cyanotic congenital heart disease, congestive heart failure, coronary artery disease; chronic respiratory conditions including suppurative lung disease, bronchiectasis, cystic fibrosis, chronic obstructive pulmonary disease, severe asthma (requiring frequent medical consultations or the use of multiple medicines); chronic neurological conditions including hereditary and degenerative CNS diseases, seizure disorders, spinal cord injuries, neuromuscular disorders; chronic metabolic disorders including Type 1 or 2 diabetes, amino acid disorders, carbohydrate disorders, cholesterol biosynthesis disorders, fatty acid oxidation defects, lactic acidosis, mitochondrial disorders, organic acid disorders, urea cycle disorders, vitamin/cofactor disorders, porphyria; chronic renal failure; children aged 5 to 10 years receiving long term aspiring therapy; Down syndrome; obesity (body mass index ≥30 kg/m2); children born less than 37 weeks gestation

Exclusion Criteria:

* COVID-19 pregnant women RCT: Pregnant women have contraindications to COVID-19 vaccines and already randomised to influenza RCT.
* Influenza pregnant women RCT: Pregnant women have contraindications to Influenza vaccines and already randomised to COVID-19 RCT.
* COVID-19 medically at risk children RCT:

  * Known contraindications to COVID-19 vaccine
  * Up to date for COVID-19 vaccine (≥ two doses) at the time of enrolment,
  * Sibling of a child already enrolled in the trial (only the sibling who is eligible and scheduled to attend a paediatric clinic first will be eligible)
  * Previous participation in the influenza nudge RCT
* Influenza medically at risk children RCT:

  * Known contraindications to influenza vaccine
  * Already received an influenza vaccine during the flu season in 2023
  * Sibling of a child already participating in the trial (the sibling who is eligible and scheduled to attend a paediatric clinic first will be eligible)
  * Previous participation in the COVID-19 nudge RCT

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1038 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of pregnant women in intervention versus standard care arm receiving one dose of the seasonal influenza vaccine, as assessed using the Australian Immunisation Register (AIR). | From the date of randomisation until the date of first documented delivery, assessed up to 42 weeks
  The difference in proportion of pregnant women in the intervention versus standard care (non-intervention) group receiving one dose of influenza vaccine from the time of randomisation during pregnancy until one month after delivery will be assessed using the vaccination status data recorded in the Australian Immunisation Register (AIR).
To determine the proportion of medically as risk children in the intervention versus standard care group receiving at least one dose of the seasonal influenza vaccine, as assessed using the Australian Immunisation Register (AIR) | Within 3 months after randomisation
  The difference in proportion of medically as risk children in the intervention versus standard care (non-intervention) group receiving at least one dose of the seasonal influenza vaccine within 3 months after randomisation will be assessed using the vaccination status data recorded in the Australian Immunisation Register (AIR).
To determine the proportion of pregnant women in intervention versus standard care arm receiving one dose of the COVID-19 vaccine, as assessed using the Australian Immunisation Register (AIR). | From the date of randomisation until the date of first documented delivery, assessed up to 42 weeks
  The difference in proportion of pregnant women in the intervention versus standard care (non-intervention) group receiving one or more doses of a COVID-19 vaccine from the time of randomisation during pregnancy until one month after delivery will be assessed using the vaccination status data recorded in the Australian Immunisation Register (AIR).
To determine the proportion of medically as risk children in the intervention versus standard care group receiving at least one dose of a COVID-19 vaccine, as assessed using the Australian Immunisation Register (AIR) | Within 3 months after randomisation
  The difference in proportion of medically at risk children receiving at least one dose of a COVID-19 vaccine within 3 months after randomisation will be assessed using the vaccination status data recorded in the Australian Immunisation Register (AIR).

SECONDARY OUTCOMES:
Number of pregnant women who received COVID-19 or influenza vaccines, change from baseline to one month post-delivery, based on socio-demographic characteristics | From the date of randomisation until one month after the date of first documented delivery, assessed up to 46 weeks
  Number of pregnant participants who received COVID-19 or influenza vaccines, change from baseline up to one month post-delivery, based on socio-demographic characteristics using the hospital records and Australian Immunisation Register (AIR).
Number of medically at risk children who received COVID-19 or influenza vaccines, change from baseline up to three months post-randomisation, based on socio-demographic characteristics | From date of randomisation until the date of first documented influenza or COVID-19 vaccination, assessed up to 3 months
  Number of medically at risk pediatric participants who received COVID-19 or influenza vaccines, change from baseline up to three months post-randomisation, based on socio-demographic characteristics using the hospital records and Australian Immunisation Register (AIR).
To assess timeliness of influenza/ COVID-19 vaccine uptake among pregnant women during the study period by determining the proportion of pregnant women who receive the influenza or COVID-19 vaccine by month throughout the study period. | From the date of randomisation until one month after the date of first documented delivery, assessed up to 46 weeks
  Timeliness of influenza and COVID-19 vaccine uptake among pregnant women during the study period will be assessed by determining the difference in proportion of pregnant women who receive the COVID-19 or influenza vaccine by month throughout the study period using the vaccination status data recorded in the Australian Immunisation Register (AIR).
To assess timeliness of influenza and COVID-19 vaccine uptake among medically at risk children during the study period by determining the proportion of medically at risk children who receive the COVID-19 or influenza vaccine by month. | From date of randomisation until the date of first documented influenza or COVID-19 vaccination, assessed up to 3 months
  Timeliness of influenza and COVID-19 vaccine uptake among medically at risk children during the study period by determining the difference in proportion of medically at risk children who receive the COVID-19 or influenza vaccine by month throughout the study period using the vaccination status data recorded in the Australian Immunisation Register (AIR).
To estimate the cost-effectiveness of proven interventions compared to standard care in hospital settings | From the date of randomisation until 46 weeks after randomisation
  The incremental cost per additional person vaccinated will be assessed by comparing interventions to standard care in hospital settings. The cost per quality-adjusted life year (QALY) gained for influenza vaccination will be assessed. Implementation costs will be obtained from the study budget and costs related to research activities will be excluded. Estimated cost offsets to the health system associated with influenza related disease (e.g. hospitalisations and emergency visits) will be derived from the literature and calculated using cost weights for Australian Refined Diagnosis Related Groups (AR-DRGs).
To determine the difference in proportion of pregnant women in intervention versus standard care arm receiving one dose of the influenza/COVID-19 vaccine, as assessed using the Australian Immunisation Register (AIR). | From the date of randomisation until one month after the date of first documented delivery, assessed up to 46 week
  The difference in proportion of pregnant women who receive one dose of influenza/COVID-19 vaccine from the time of randomisation during pregnancy until one month after delivery will be assessed using the vaccination status data recorded in the Australian Immunisation Register (AIR).

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Women's and Children's Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Mercy Hospital For Women, Heidelberg, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia
  - King Edward Memorial Hospital, Subiaco, Western Australia

REFERENCES:
- [Derived] Wang B, Andraweera P, Danchin M, Blyth CC, Vlaev I, Ong J, Dodd JM, Couper J, Sullivan TR, Karnon J, Spurrier N, Cusack M, Mordaunt D, Simatos D, Dekker G, Carlson S, Tuckerman J, Wood N, Whop LJ, Marshall H. Nudging towards COVID-19 and influenza vaccination uptake in medically at-risk children: EPIC study protocol of randomised controlled trials in Australian paediatric outpatient clinics. BMJ Open. 2024 Feb 17;14(2):e076194. doi: 10.1136/bmjopen-2023-076194. PMID 38367966
- [Derived] Andraweera PH, Wang B, Danchin M, Blyth C, Vlaev I, Ong J, Dodd J, Couper J, Sullivan TR, Karnon J, Spurrier N, Cusack M, Mordaunt D, Simatos D, Dekker G, Carlson S, Tuckerman J, Wood N, Whop L, Marshall HS. Randomised controlled trials of behavioural nudges delivered through text messages to increase influenza and COVID-19 vaccines among pregnant women (the EPIC study): study protocol. Trials. 2023 Jul 12;24(1):454. doi: 10.1186/s13063-023-07485-9. PMID 37438776